CLINICAL TRIAL: NCT03778190
Title: The Use of a Magnet to Remove Corneal Foreign Bodies
Brief Title: Magnet for Corneal Foreign Bodies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kendall Healthcare Group, Ltd. (Industry)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018-419-Non-NSU Health
Record Dates: First submitted 2018-12-14; First posted 2018-12-19 (Actual); Results first posted 2020-08-26 (Actual); Last update posted 2020-08-26 (Actual); Status verified 2020-08

CONDITIONS: Corneal Foreign Body

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Magnet (Experimental): The physician will attempt to remove the corneal foreign body using an eye magnet for these patients.
  Interventions: Procedure: Corneal Foreign Body Removal

INTERVENTIONS:
Procedure: Corneal Foreign Body Removal — An eye magnet will be brought close to the foreign body on the surface of the eye in an attempt to remove the foreign body.

SUMMARY:
This is a prospective, interventional study to assess the effectiveness and safety of a commercially available "eye magnet" to remove corneal foreign bodies.

DETAILED DESCRIPTION:
The vast majority of corneal foreign bodies are metallic and thus are frequently ferromagnetic. Consequently, it may be possible to use a magnet to remove most corneal foreign bodies. There are commercially available products for removing corneal foreign bodies, but there are no published studies assessing these devices.

This will be a prospective interventional study to assess the use of an eye magnet for the removal of metallic corneal foreign bodies in the emergency department.

After the patient signs written, informed consent, the physician will attempt to remove the corneal foreign body with the North by Honeywell 326734G Eye Magnet with Loop. If the physician is unable to remove the corneal foreign body with the magnet, he or she may proceed with standard care.

The treating physician will fill out a brief data collection form for each patient to track various outcomes as discussed below.

ELIGIBILITY:
Inclusion Criteria:

* present to the emergency department with a metallic corneal foreign body

Exclusion Criteria:

* prisoners
* pregnant women
* have pacemakers or metallic facial implants
* possible globe rupture

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-12-04 (Actual); Primary Completion 2019-11-11 (Actual); Study Completion 2019-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tony Zitek, MD, Study Director — Kendall Healthcare Group, Ltd.
Locations (1):
- Kendall Regional Medical Center, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Magnet
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Magnet
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: The percentage of patients in whom the magnet successfully removed the foreign body.
Time Frame: 5 minutes.
Measure: Count of Participants; unit: Participants
Arm/Group | Magnet
Number analyzed (Participants) | 10
Participants | 1

2. Secondary Outcome: Epithelial Damage
Description: The percentage of patients in whom the amount of fluorescein uptake on exam was more after the procedure compared to before the procedure.
Time Frame: 5 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Magnet
Number analyzed (Participants) | 10
Participants | 0

ADVERSE EVENTS:
Time Frame: 10 minutes
Arm/Group | Magnet
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 0/10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/90/NCT03778190/Prot_000.pdf